CLINICAL TRIAL: NCT06587048
Title: Outcome of Bone Window Approach in Endodontic Microsurgery Using Novel Piezoelectric Device Versus Conventional Rotary Burs in the Treatment of Periapical Lesions - a Randomized Controlled Trial
Brief Title: Outcome of Bone Window Approach in Endodontic Microsurgery Using Novel Piezoelectric Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, principal investigator, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: keerthana
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Periapical Lesions; Chronic Apical Periodontitis of Pulpal Origin
Keywords: endondontic microsurgery; piezoelectric device; piezoendodontic surgery; bone window

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Piezo group (Experimental): The bone window osteotomy will be created with a piezoelectric device during endodontic microsurgery
  Interventions: Procedure: periapical surgery
- conventional bur group (Active Comparator): The bone window osteotomy will be created with a conventional rotary burs in slow-speed handpiece during endodontic microsurgery
  Interventions: Procedure: periapical surgery

INTERVENTIONS:
Procedure: periapical surgery — In piezo group, the periapical surgery will be performed using piezoelectric device.
  Arms: Piezo group
Procedure: periapical surgery — In conventional bur group, the periapical surgery will be performed using rotary burs.
  Arms: conventional bur group

SUMMARY:
The Bone window technique provides excellent access to the surgical site while preserving cortical bone in cases of tooth with large periapical lesion and an intact cortical plate. Traditionally, rotary burs and a bone chisel were used to create a bone window. Piezoelectric bone surgery, on the other hand, is an innovative technique that uses thin osteotomy instrument to selectively cut hard tissue while preserving soft tissues. To the best of our knowledge, no study comparing the results of a bone lid using a piezoelectric device and a conventional bur is currently available.

DETAILED DESCRIPTION:
Endodontic microsurgery is the treatment option frequently opted to manage endodontically failed cases with persistent apical periodontitis, after nonsurgical root canal treatment (1,2). Contemporary surgical endodontic therapy using dental operating microscope enables a more precise technique with no or little bevel of root-end excision and retrograde canal preparation with an ultrasonic tip to a depth of 3-4 mm (3). The cumulative loss of cortical bone may further result in slowed or unsuccessful healing at the surgical site as a result of the disease process and/or the removal of cortical plates during a surgical procedure (4,5). According to the animal histologic sections, the cortical plate heals slowest, with a 70% healing rate at the 6-month follow-up. Von Arx et al reported that only 54.1% of patients demonstrated complete cortical plate healing at the end of one-year follow-up when assessed by cone-beam computed tomography (CBCT) (6). The degree of cortical plate loss and its limited capacity for regeneration may necessitate the use of regenerative methods involving graft materials.

A novel and minimally invasive procedure called the bone window approach to the apical region aims to preserve more bony structure and the structural integrity of the healthy cortical plate. The bone window also functions as autologous graft material, which has been recognized as the gold standard for regeneration without the need for additional substitute materials (7,8). For obtaining bone window, use of traditional burs in combination with chisels, reciprocating or oscillating saws and lasers have been reported in literature. Piezoelectric bone surgery is an innovative technology that has gained popularity in recent years. It makes use of thin osteotomy instruments that enable selective hard tissue cutting while safeguarding soft tissues (9). This technique is not only clinically effective, but histological and histomorphometric evidence of wound healing and bone formation in experimental animal models has shown that tissue response is better in piezo surgery than in conventional bone-cutting techniques such as diamond or carbide rotary instruments (10-12).

In cases of large periapical lesions where the buccal cortical plate is intact, the application of the piezoelectric device has recently been reported in case reports to create a bony window on buccal bone (13, 14). In a recent randomized trial (15), piezo surgery was compared to traditional microsurgery to assess haemorrhage control and patient postoperative quality of life. In a recent randomized trial (16) comparing bone lid technique over traditional technique in the surgical management of mandibular lesions, the bone lid technique using a piezoelectric device was found to be safe and effective for treating lesions in the posterior mandibular region and was associated with less postoperative complications. The bone lid approach has been used in the literature on oral and maxillofacial surgery for a number of procedures, including root-end surgery, cystic enucleation, impacted tooth extraction, implant explantation, and access to the maxillary sinus for the removal of cysts or foreign bodies. The review concluded that the included clinical studies were of low quality evidence, and that randomized clinical trials were necessary to compare the effectiveness of the bone lid technique to other methods. Furthermore, the best cutting tool for fashioning bone lids has not yet been identified (17).

The transition of endodontic diagnosis and treatment planning from two dimensions to three dimensions is facilitated by CBCT scanning, which also shows the location of anatomical structures in three dimensions, provides precise measurements in depth and length, and enhances localization of the periapical lesion (18, 19). Furthermore, CBCT imaging has high sensitivity to detect the presence of a bony defect in the cortical plate and precisely measure its thickness (20, 21, 22).

ELIGIBILITY:
Inclusion Criteria:

* • Consenting adults (age range: 18-60 years)

  * Non-contributory medical history (ASA Class I or Class 2)
  * Participants with symptomatic/persistent apical periodontitis showing clinical signs and symptoms and evidence of periapical lesion of strictly endodontic origin with minimum lesion diameter of 5mm on periapical radiography (PR).
  * Radiographic evidence of an intact buccal cortical plate on cone-beam computed tomographic (CBCT) imaging with minimum thickness of 1mm.

Exclusion Criteria:

* Patients with systemic diseases (diabetes mellitus, uncontrolled hypertension, hepatic/renal disease, or systemic bleeding disorders), pregnancy, smoking
* Patients on anticoagulant/ antiplatelet drugs
* Teeth that were unrestorable, fractured/perforated teeth,
* Teeth with endodontic-periodontal communication and
* Teeth with deep pockets (probing depth >4 mm)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
clinical assessment | 1 year after surgery
  All patients will undergo surgical evaluation 24 h, 48h, 72 h, one week, six months and 12 months after the surgery. Postsurgical pain was measured using the VAS scale.
Radiographic outcome | 1 year after surgery
  CBCT will be performed 12 months postoperatively, and the findings will be compared with preoperative CBCT findings to assess the bone defect fill and cortical plate formation using modified PENN 3D criteria and RAC index

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India